CLINICAL TRIAL: NCT04392297
Title: To Identify the Clinical and Immunological Features of the CMV Infection Atypical Course in Immunocompetent Individuals and to Develop Methods for the Diagnosis and Treatment of Patients in This Category
Brief Title: Clinical and Immunological Features of the CMV Infection Atypical Course in Immunocompetent Individuals
Status: Completed | Type: Observational
Sponsor: The Republican Research and Practical Center for Epidemiology and Microbiology (Other)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: RRPCEM_CMV
Record Dates: First submitted 2020-05-11; First posted 2020-05-18 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: CMV
Keywords: Cytomegalovirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Heparinized whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CMV infection
  Interventions: Diagnostic Test: Bood leukocyte subsets; Diagnostic Test: CMV specific T-cells; Diagnostic Test: serum CMV IgM / IgG antibodies

INTERVENTIONS:
Diagnostic Test: Bood leukocyte subsets — Determination of blood leukocyte subpopulations: myeloid suppressor cells, T-regulatory cells, T-cells according to the stages of differentiation (naive - effector - memory), activated T-cells; circulating endothelial cells
Diagnostic Test: CMV specific T-cells — CMV specific T-cells detected by flow cytometry
Diagnostic Test: serum CMV IgM / IgG antibodies — serum CMV IgM / IgG antibodies detected by ELISA

SUMMARY:
Current study evaluates possible correlations between the content of various cell populations, the genetic material of the virus and antibodies to it in the blood of patients and the risk of thrombosis development in patients with acute CMV infection.

А new method for the early detection of immunological and clinical signs of thromboembolic complications of CMV infection in immunocompetent individuals and the treatment of patients in this category will be developed.

DETAILED DESCRIPTION:
* evaluate the immune status main indicators that characterize the activation of immune system, immunosuppression and anergy (myeloid suppressor cells, T-regulatory cells, T-cells according to the stages of differentiation (naive - effector - memory), activated T-cells);
* identify and characterize immunological disorders in patients with CMV infection complicated by thromboembolism of various localization;
* determine the presence and quantitative content in plasma / serum and neutrophils of the CMV genetic material by real-time PCR;
* study humoral immunity to CMV (IgM / IgG antibodies to CMV in serum);
* determine the content of CMV specific T-cells in peripheral blood;
* develop a method for the early detection of immunological and clinical signs of thromboembolic complications of CMV infection in immunocompetent persons and treatment of patients in this category.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 80 years;
* fever of not clear etiology
* confirmed CMV infection

Exclusion Criteria:

* HIV infection
* taking hormones, cytostatics;
* drug addiction
* malignant neoplasms over the past 5 years.
* active viral hepatitis or liver cirrhosis;
* immunosuppressive conditions of any etiology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with CMV infection
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with thrombosis | 1 month
  Thrombosis as a complication of CMV infection and its association with immune status, CMV specific T-cells count and CMV specific antibodies level

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fomina, Dr, Principal Investigator — Head of the laboratory, RSPCEM
Locations (1):
- The Republican Research and Practical Center for Epidemiology and Microbiology, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No